CLINICAL TRIAL: NCT01831557
Title: The Genetic Basis of the Influence of Dairy Product Intake on Body Measures in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-18-2012
Record Dates: First submitted 2013-04-04; First posted 2013-04-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Body Mass Index
MeSH Terms: interventions — Base Sequence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Childrens' Milk Intake: The milk intake of children will be reconciled with body measurement index and blood samples will be taken for gene sequencing
  Interventions: Other: Blood samples will be taken for gene sequencing

INTERVENTIONS:
Other: Blood samples will be taken for gene sequencing

SUMMARY:
The objective of this study is to explore the genetic basis of the influence of dairy product intake on body measures in children. The investigators assume that the effect of dairy products intake on children body measures is affected by genetic polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children

Exclusion Criteria:

* Sick children
* Chronic diseases

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children from a community sample
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Body indexes measurements | One year
  Body indexes measurements including height and weight in correlation with milk intake and gene sequences.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel